CLINICAL TRIAL: NCT02682758
Title: Influence of Xenon Anaesthesia on Transpulmonary Pressure and Tidal Volume Distribution
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 5161R
Record Dates: First submitted 2016-02-04; First posted 2016-02-15 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Anesthesia
Keywords: xenon; transpulmonary pressure; electrical impedance tomography; tidal volume; esophageal pressure measurement
MeSH Terms: interventions — Xenon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients of normal weight (Other): Patients undergoing routine xenon-based general anaesthesia for surgery with a body mass index of less than 30.
  Interventions: Drug: Xenon
- Obese patients (Other): Patients undergoing routine xenon-based general anaesthesia for surgery with a body mass index equal to or more than 30.
  Interventions: Drug: Xenon

INTERVENTIONS:
Drug: Xenon — Wash-in of xenon for maintenance of anaesthesia
  Other Names: Xenon pro Anaesthesia

SUMMARY:
The influence of xenon anaesthesia on transpulmonary pressure and tidal volume distribution will be investigated in a prospective cohort study in 10 patients of normal weight and 10 obese patients undergoing routine xenon-based, general anaesthesia for surgery.

DETAILED DESCRIPTION:
To investigate the influence of xenon-anaesthesia on transpulmonary pressure and tidal volume Distribution, the investigators will enroll 20 patients - 10 with a Body mass index of less than 30 and 10 with a Body mass index of 30 or more - undergoing routine xenon-based anesthesia in the course of a prospective cohort study. Performance of anesthesia will be at the discretion of the attending anesthesiologist. Typically, xenon-based anesthesia is induced and initially maintained with propofol and an opioid and tracheal intubation is facilitated using a muscle relaxant. Initially, the patient is ventilated with 100 per cent oxygen in order to wash out nitrogen from the respirator and the lungs. When nitrogen wash-out is completed, 55-65 per cent xenon in oxygen is introduced.

5 minutes after anaesthesia induction, as well as 5 minutes after completion of Xenon wash-in, transpulmonary pressure will be measured from inspiratory plateau pressure and pleural pressure, which will be estimated from esophageal pressure. Esophageal pressure measurements will be facilitated via esophageal balloon catheters (Adult Esophageal Balloon Catheter Set 5 French, CooperSurgical, Trumbull, USA).

Tidal volume distribution will be assessed with the use of Electrical Impedance Tomography (EIT). Images will be acquired in the supine Position 5 minutes before anesthesia induction, 5 minutes after induction as well as 5 minutes completion of xenon wash-in. EIT measurements will be made for a period of one minute and functional EIT images of changes in tidal impedance will be generated. The Center of Ventilation Index and Global Inhomogeneity Index will be calculated for each time point.

Analysis Plan:

The primary analysis will include all recruited patients, irrespective of their Body mass index. Changes in transpulmonary pressure before and after Xenon wash-in will be assessed with the Wilcoxon signed-rank test for matched pairs. Center of Ventilation Index and Global Inhomogeneity Index, which will be assessed at three time points, will be compared with the use of repeated measures ANOVA with the post-hoc Sidak test.

Secondary subgroup analyses will consist of separate analyses for patients with a BMI over or equal to and a BMI of less than 30. A type I error will be accepted with a maximum probability of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* Xenon-based, general anaesthesia for elective surgery independent of this investigation

Exclusion Criteria:

* Inability to provide informed consent
* Known pregnancy
* American Society of Anesthesiologists status >III
* Restrictive or obstructive pulmonary disease
* History of esophageal or gastric operation
* Esophageal varices
* Liver cirrhosis Child-Pugh B or C
* Therapeutic anticoagulation
* Cardiac pacemaker or internal automatic defibrillator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in transpulmonary pressure after Xenon wash-in | 5 minutes before and 5 minutes after xenon-wash in

SECONDARY OUTCOMES:
Change in tidal volume Distribution as measured by Electrical impedance tomography | 5 minutes before induction of anaesthesia, 5 minutes before 5 minutes after xenon wash-in

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kienbaum, MD, Principal Investigator — Klinik für Anästhesiologie, Universitätsklinikum Düsseldorf, Germany
Locations (1):
- Department of Anesthesiology, Düsseldorf University Hospital, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Frerichs I, Dargaville PA, van Genderingen H, Morel DR, Rimensberger PC. Lung volume recruitment after surfactant administration modifies spatial distribution of ventilation. Am J Respir Crit Care Med. 2006 Oct 1;174(7):772-9. doi: 10.1164/rccm.200512-1942OC. Epub 2006 Jul 13. PMID 16840739
- [Background] Zhao Z, Moller K, Steinmann D, Frerichs I, Guttmann J. Evaluation of an electrical impedance tomography-based Global Inhomogeneity Index for pulmonary ventilation distribution. Intensive Care Med. 2009 Nov;35(11):1900-6. doi: 10.1007/s00134-009-1589-y. Epub 2009 Aug 4. PMID 19652949
- [Derived] Schaefer MS, Treschan TA, Gauch J, Neukirchen M, Kienbaum P. Influence of xenon on pulmonary mechanics and lung aeration in patients with healthy lungs. Br J Anaesth. 2018 Jun;120(6):1394-1400. doi: 10.1016/j.bja.2018.02.064. Epub 2018 Apr 13. PMID 29793604